CLINICAL TRIAL: NCT05572541
Title: Assessment of Temporomandibular Joint Dysfunction in Patients With Traumatic Brain Injury
Brief Title: Temporomandibular Joint Dysfunction in Patients With Traumatic Brain Injury
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Konya Beyhekim Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Savaş Karpuz, Medical doctor, Konya Beyhekim Training and Research Hospital
Other Study IDs: 2022-01-04
Record Dates: First submitted 2022-10-04; First posted 2022-10-07 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Temporomandibular Dysfunction
Keywords: Temporomandibular Dysfunction,; traumatic brain injury; headache
MeSH Terms: conditions — Temporomandibular Joint Disorders; Brain Injuries, Traumatic; Headache

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with traumatic brain injury: Temporomandibular joint range of motion, Fonseca questionnaire, facial asymmetry, and massater and temporal pain threshold will be evaluated by measuring both TBI patients and healthy individuals. In addition, post-injury dietary intake and dominant chewing side will be questioned in TBI patients. Temporomandibular movements will be measured with a disposable cardboard ruler.
  Interventions: Diagnostic Test: Fonseca questionnaire
- healthy volunteers: Temporomandibular joint range of motion, Fonseca questionnaire, facial asymmetry, and massater and temporal pain threshold will be evaluated by measuring both TBI patients and healthy individuals. Temporomandibular movements will be measured with a disposable cardboard ruler.
  Interventions: Diagnostic Test: Fonseca questionnaire

INTERVENTIONS:
Diagnostic Test: Fonseca questionnaire — Fonseca questionnaire for the evaluation of temporomandibular dysfunction
  Other Names: Joint range of motion measurement,; pressure pain threshold measurement

SUMMARY:
Trauma, neurological disorders and psychological problems, which are the etiological factors of temporomandibular joint dysfunction, can be seen in patients with traumatic brain injury.

The aim of this study is to investigate temporomandibular joint dysfunction in patients with traumatic brain injury.

Participants (traumatic brain injury patients and healthy volunteers) will be evaluated once for temporomandibular joint dysfunction.

DETAILED DESCRIPTION:
Temporomandibular joint range of motion, Fonseca questionnaire, facial asymmetry, and massater and temporal pain threshold will be evaluated by measuring both TBI patients and healthy individuals. In addition, post-injury dietary intake and dominant chewing side will be questioned in TBI patients. Temporomandibular movements will be measured with a disposable cardboard ruler.

Exclusion criteria; communication and cooperation problems, congenital or systemic disease affecting the head and neck region, being treated for TMED and having a history of orthognathic surgery.

ELIGIBILITY:
Inclusion Criteria:

clinical diagnosis of traumatic brain injury not receiving treatment for temporomandibular joint dysfunction

Exclusion Criteria:

communication and cooperation problems, congenital or systemic disease affecting the head and neck region, being treated for TMED and having a history of orthognathic surgery.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 30 Patient with traumatic brain injury 30 healthy volunteer
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-11-05 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of temporomandibular joint dysfunction in patients with traumatic brain injury | 01.11.2022

CONTACTS AND LOCATIONS:
Locations (1):
- Konya Beyhekim Research and Training Hospital, Konya, Selçuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
We will share if requested.